CLINICAL TRIAL: NCT07258862
Title: Analysis of Microbial Biofilms in Peripheral Venous Catheters and Their Implication in Infectious Risk
Acronym: KTBIO
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital NOVO (Other)
Collaborators: Université de Cergy Pontoise (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHRD1025; 202509 - 011 (Other: Université Cergy Pontoise)
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Catheter-Related Infections
Keywords: Vascular Access Devices; Peripheral Venous Catheter; Catheter-Related Infections; Biofilms; Molecular Biology; Next-Generation Sequencing; Scanning Electron Microscopy
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inflammatory catheters: Catheter removed because of infection at insertion site
  Interventions: Diagnostic Test: Inflammatory catheters: catheter removed because of infection at insertion site
- Non-inflammatory catheters: catheter removed because it is no longer relevant to keep it in place
  Interventions: Device: Non-inflammatory catheters: catheter removed because it is no longer relevant to keep it in place

INTERVENTIONS:
Diagnostic Test: Inflammatory catheters: catheter removed because of infection at insertion site — Verification of inclusion and non-inclusion criteria (at least 2 days and at most 7 days, with or without signs of inflammation).
  The doctor or a qualified nurse orally informs the patient when catheter removal is planned.
  The information and non-opposition note are given to the patient, and the information procedure is recorded in the medical record.
  The catheter is removed and collected under aseptic conditions by the nurses in the various departments, in a dry sterile tube. The tube is then labelled and stored at a maximum of 4°C. The catheter is sent to the hospital's biology laboratory before being collected by the approved carrier for delivery to the ERRMECe laboratory from CYU. All tests are performed in the ERRMECe laboratory. Collected catheters are subsequently analysed to assess the bacterial diversity of biofilms using molecular biology techniques and Next-Generation Sequencing (NGS), in parallel with biofilm structural analysis microscopy using a Scanning Electron Microsc
  Groups: Inflammatory catheters
Device: Non-inflammatory catheters: catheter removed because it is no longer relevant to keep it in place — Verification of inclusion and non-inclusion criteria (at least 2 days and at most 7 days, with or without signs of inflammation).
  The doctor or a qualified nurse orally informs the patient when catheter removal is planned.
  The information and non-opposition note are given to the patient, and the information procedure is recorded in the medical record.
  The catheter is removed and collected under aseptic conditions by the nurses in the various departments, in a dry sterile tube. The tube is then labelled and stored at a maximum of 4°C. The catheter is sent to the hospital's biology laboratory before being collected by the approved carrier for delivery to the ERRMECe laboratory from CYU. All tests are performed in the ERRMECe laboratory. Collected catheters are subsequently analysed to assess the bacterial diversity of biofilms using molecular biology techniques and Next-Generation Sequencing (NGS), in parallel with biofilm structural analysis microscopy using a Scanning Electron Microsc
  Groups: Non-inflammatory catheters

SUMMARY:
Peripheral venous catheters (PVCs) are the most commonly used intravascular medical devices in healthcare establishments. Although essential in patient care, PVCs represent a significant risk factor for nosocomial infections, as shown by the results of the national prevalence survey. While the main pathophysiological mechanisms are known, the specific factors driving the transition from simple colonization to infection remain unclear. This project aims to identify the major factors involved in the occurrence of bacterial infections related to the colonization of peripheral venous catheters.

DETAILED DESCRIPTION:
Peripheral venous catheters (PVCs) are the most commonly used intravascular medical devices in healthcare establishments. In the 2022 national survey on the prevalence of nosocomial infections (NI), out of 151676 patients included, 22.45% had a peripheral venous catheter. Moreover, patients exposed to a PVC are 3 times more likely to suffer a nosocomial infection. Between 2019 and 2023, at national level, there was a significant increase in the proportion of PVC-related bloodstream infection. The pathophysiological mechanisms of catheter-related infections are mainly linked to contamination via the endoluminal route, through manipulations of connectors during perfusion connections, or via the extraluminal route, which is more likely to be associated with faulty catheter placement practices. Finally, even in patients with no clinical signs of infection, culture-negative PVCs show intra- and extra-luminal colonization.

This underscores our lack of understanding of the mechanisms that can lead from simple colonization of the equipment to localized catheter infection or even bacteraemia.

The main objective of this project is to identify the major factors involved in the occurrence of bacterial infections related to the colonization of peripheral venous catheters.

To investigate these mechanisms, the study will focus on the collection of PVCs after clinical removal, followed by molecular and super-resolution microscopy analyses. Catheters either removed by the care team, because they are no longer clinically relevant or for medical reasons, will be collected under aseptic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in a care unit of the NOVO hospital (Pontoise site)
* Major patient for whom a peripheral venous catheter has been in place for at least 2 days and at most 7 days, with or without signs of inflammation

Exclusion Criteria:

* Antibiotic treatment by any route
* Patient with viral hepatitis, or human immunodeficiency virus (HIV) or suspected epidemic and biological risk (EBR)
* Patient unable to understand and give non-opposition to study participation
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in a care unit of the NOVO hospital
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Bacterial diversity of biofilms in PVCs according to inflammatory symptoms | 15 months
  Relative abundance of bacteria within biofilms present in CVPs as identified by NGS, according to inflammatory symptoms.

SECONDARY OUTCOMES:
Biofilms structural morphology in PVCs | 15 months
  Qualitative imaging of microbial biofilms in PVCs using Scanning Electron Microscopy
Bacterial diversity of biofilms in PVCs according to type of substances administered through the vascular route | 15 months
  Relative abundance of bacteria within biofilms present in PVCs as identified by NGS, according to the type of substances received by patients through the vascular route
Bacterial diversity of biofilms in PVCs according to catheter dwell time | 15 months
  Relative abundance of bacteria within biofilms present in CVPs as identified by NGS, according to catheter dwell time.

CONTACTS AND LOCATIONS:
Overall Officials: LECURU Marion, Doctor, Principal Investigator — Hôpital NOVO
Locations (2):
- France (2):
  - Hopital Novo, Cergy-Pontoise, Hopital NOVO
  - CY Cergy Paris Université, Neuville-sur-Oise

IPD SHARING:
Plan to Share IPD: No